CLINICAL TRIAL: NCT04807829
Title: A Randomized-Controlled Trial With the Adjunctive CB1 Agonist Nabilone in Inpatients With Active Suicidal Ideation
Brief Title: Adjunctive CB1 Agonist Nabilone in Inpatients With Active Suicidal Ideation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to drug unavailability. The drug is unavailable because production was discontinued in the US.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rodrigo Machado-Vieira, MD, PhD, MSc, Professor of Psychiatry, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-20-1312
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nabilone (Experimental): Patients in the treatment group will be administered oral Nabilone 2 mg once daily for 3 days in addition to treatment as usual according to current clinical guidelines and standard of care.
  Interventions: Drug: Nabilone
- Placebo Comparator (Placebo Comparator): Patients in the Placebo Comparator group will receive placebo once daily for 3 days plus treatment as usual.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Nabilone is a synthetic endocannabinoid and CB1 agonist.
  Other Names: Cesamet
  Arms: Nabilone
Drug: Placebo — Inactive placebo comparator
  Arms: Placebo Comparator

SUMMARY:
Suicide is a major crisis worldwide with rates projected to continue to increase. There is currently a dearth of novel pharmacologic treatment options for suicide available on the market. The endocannabinoid system has been recently shown to be associated with mood disorders including suicidality. The aim of the study is to determine whether treatment with Nabilone is capable of reducing suicidal ideation in adults after 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Current suicidal ideation
* Columbia Suicide Severity Rating Scale (CSSRS) score of ≥ 4 and Scale for Suicide Ideation (SSI) first 5 items, score of ≥4
* Current major depressive episode as evidenced by MADRS score ≥ 20

Exclusion Criteria:

* Current diagnosis of a Diagnostic and Statistical Manual V (DSM-V) psychotic disorder, psychotic symptoms, or personality disorder.
* Recent (<72 hrs) use of illicit substances
* Comorbid substance use disorder diagnosis
* Urine drug screen (UDS) positive for tetrahydrocannabinol (THC)
* Pregnant or nursing women
* Unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal Ideation and Behavior as assessed by an abbreviated version of the Columbia-Suicide Severity Rating Scale (CSSRS) | baseline, day 3
  For the abbreviated, six-question version of the CSSRS, total scores range from 0 to 6 with a higher score indicating greater suicidal ideation and behavior.

SECONDARY OUTCOMES:
Change in Depression as assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) | baseline, day 3
  The MADRS is a ten item instrument, with each of the ten items rated on a scale of 0 to 6, giving a total score range of 0 to 60. A higher score indicates greater depression.
Change in Suicidal Ideation as assessed by the Scale for Suicide Ideation (SSI) | baseline, day 3
  The SSI is a nineteen item measure of current suicidal ideation and intention, with each item rated on a scale of 0 to 2, giving a total score range of 0 to 38. A higher score indicates greater suicidal ideation and intention.
Change in Anxiety as assessed by the General Anxiety Disorder-7 (GAD-7) | baseline, day 3
  The GAD-7 is a seven item instrument, with each of the 7 items is scored from 0 to 3, giving a total score range of 0 to 21. A higher score indicates greater anxiety.

OTHER OUTCOMES:
Biomarkers | baseline, day 3
  To determine whether treatment with Nabilone would lead to changes in the level of serum biomarkers and inflammatory cytokines; and their association with its antisuicidal and antidepressant effects.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Machado-Vieira, MD, PhD, MSc, Principal Investigator — UTHealth
Locations (1):
- Harris County Psychiatric Center (HCPC), Houston, Texas, United States